CLINICAL TRIAL: NCT05287997
Title: A 2-Part Capillary Blood Biomarker Cohort Study to Diagnose Adolescent Sport Concussion
Brief Title: Blood Biomarker Study to Diagnose Adolescent Sport Concussion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neurolytixs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NLI01
Record Dates: First submitted 2022-02-22; First posted 2022-03-18 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Participants will enrol into the Baseline Arm of the study. Participants will attend all Baseline Visits unless they experience a concussion at which point, they will transition to the Concussion Arm for further follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (Other): Participants in this arm will be evaluated at 3 time periods. Initial pre-season visit, mid-season visit and end-of-season visit. Capillary blood sample collection will occur at each visit.
  Interventions: Diagnostic Test: Neurolytixs Index
- Concussion (Experimental): Participants in this arm will transition from the baseline arm to the concussion arm if they experience a concussion during the course of the sporting season. They will be evaluated with 72 hours of the injury and then at 2-, 4-, and 12-weeks post-injury. Capillary blood sample collection will occur at each visit.
  Interventions: Diagnostic Test: Neurolytixs Index

INTERVENTIONS:
Diagnostic Test: Neurolytixs Index — Capillary blood sample will be collected on a dried plasma sample (DPS) filter paper. The sample will be sent to a central laboratory where they will undergo metabolite extraction and analysis via mass spectrometry.

SUMMARY:
Concussions are one of the most complex conditions to manage in sport medicine due to the individualized clinical presentation, caused by a complex neurometabolic cascade, and the lack of a diagnostic standard. There is currently no objective measurement for concussion and the reliance on subjective reporting and clinical judgement is imperfect.

In previous clinical studies the investigators determined cutoff values of plasma phosphatidylcholines that provided strong indication that a concussion had occurred. Based on this data, the investigators have developed a custom assay, which will work together with a capillary blood collection device. The current clinical trial will be conducted in two parts. Part A will allow the investigators to determine precise AUC cut-off values for the propriety, novel custom assay, and in Part B the investigators will assess the safety and efficacy of this device for concussion diagnosis in adolescent athletes aged 13-17.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent/assent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female athletes, aged 13-17 inclusive

Exclusion Criteria:

1. Individuals who have suffered a known concussion within the 6 months prior to enrollment
2. Individuals who suffer from an acute neurological disorder
3. Known pregnancy

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Part A: Calculate population reference ranges for 10 phosphatidylcholines (PC) specific to Neurolytixs assay kit. | End of Part A (4-6 months)
  Population reference values will be determined with the standard definition of a reference range as the interval between which 95% of values of a reference population fall into, in such a way that 2.5% of the time a value will be less than the lower limit of this interval, and 2.5% of the time it will be larger than the upper limit of this interval, whatever the distribution of these values. Measured PC values will be plotted against both sex and the age of participants to which the PCs were measured.
Part A: Generate Area Under the Curve (AUC) values specific to the Neurolytixs assay kit | End of Part A (4-6 months)
  Generate AUC values for 10 phosphatidylcholines (PCs) for use in Part B
Part B: Determine efficacy of Neurolytixs assay kit for diagnosing adolescent sports concussion | 12-72 hours post-injury
  The change of at least 1 PC below the cutoff threshold (determined in Part A)
Part B: Determine safety of the Neurolytixs assay kit for adolescent sports concussion | Through study completion, up to 1 year
  Calculate the number of false negatives (concussions that are not captured by the assay
Part B: Determine safety of the Neurolytixs assay kit for adolescent sports concussion | Through study completion, up to 1 year
  Calculate the number of false positives identified by the assay

SECONDARY OUTCOMES:
Part B: Determine whether repeated plasma PC measurements over time correlate with injury symptom resolution or clinical recovery | 12 weeks post-injury
  Sensitivity and specificity of the assay compared to diagnosis via the SCAT5

OTHER OUTCOMES:
Part B: Compare proportion of males and females with a change in PC1 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Part B: Compare proportion of males and females with a change in PC2 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Part B: Compare proportion of males and females with a change in PC3 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Part B: Compare proportion of males and females with a change in PC4 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Part B: Compare proportion of males and females with a change in PC5 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Part B: Compare proportion of males and females with a change in PC6 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Part B: Compare proportion of males and females with a change in PC7 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Part B: Compare proportion of males and females with a change in PC8 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Part B: Compare proportion of males and females with a change in PC9 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Part B: Compare proportion of males and females with a change in PC10 | 12 weeks post-injury
  Comparison between proportions of sexes diagnosed with concussion and their corresponding PC levels
Number of Unanticipated Adverse Device Effects | Through study completion, up to 1 year
  Frequency of UADEs

CONTACTS AND LOCATIONS:
Overall Officials: Douglas D Fraser, MD/PhD, Principal Investigator — Neurolytixs
Locations (2):
- Legacy Center Sports Complex, Brighton, Michigan, United States
- The Hill Academy, Caledon, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided